CLINICAL TRIAL: NCT05483868
Title: A Phase 1, Open-label Trial of Belzupacap Sarotalocan (AU-011) to Determine the Feasibility and Safety of Intratumoral Injection With or Without Intramural Injection in Subjects With Bladder Cancer
Brief Title: A Phase 1, Open-label Trial of Belzupacap Sarotalocan (AU-011) in Bladder Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aura Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AU-011-102
Record Dates: First submitted 2022-07-20; First posted 2022-08-02 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Non-muscle-invasive Bladder Cancer; Non-Muscle Invasive Bladder Cancer (&Amp;#34;NMIBC&Amp;#34;) Unresponsive/Intolerant to BCG; NMIBC; Non-Muscle Invasive Bladder Carcinoma; Non-Muscle Invasive Bladder Neoplasms; Non-Muscle Invasive Bladder Urothelial Carcinoma; Urothelial Carcinoma Bladder
Keywords: NMIBC; TURBT; Intramural; AU-011; Belzupacap Sarotalocan; Intratumoral; urothelial; bladder cancer; bel-sar
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (10):
- Focal injections of AU-011 prior to TURBT (1b) (Experimental): Intratumoral (50 μg) and intramural (50 μg) injection of AU-011 prior to the standard of care (TURBT) in patients with NMIBC.
  Interventions: Drug: AU-011
- Focal injections of AU-011 with laser application before TURBT (4a) (Experimental): Intratumoral (50 μg) and intramural (50 μg) injection of AU-011 with laser application before standard of care (TURBT) in patients with NMIBC.
  Interventions: Combination Product: AU-011 in Combination with Medical Laser Adminstration
- Focal injection of AU-011 with laser application before TURBT (4b) (Experimental): Focal injection of AU-011 (100 μg) with laser application before standard of care (TURBT) in patients with NMIBC.
  Interventions: Combination Product: AU-011 in Combination with Medical Laser Administration
- Focal injection of AU-011 with laser application before TURBT (4c) (Experimental): Focal injection of AU-011 (200 μg) with laser application before standard of care (TURBT) in patients with NMIBC.
  Interventions: Combination Product: AU-011 in Combination with Medical Laser Administration
- Focal injection of AU-011 and laser application with option for TURBT (4d) (Experimental): Participants with intermediate-risk NMIBC will receive multiple treatment cycles of focal AU-011 (200 ug per lesion) with laser treatment and option for TURBT in patients with intermediate risk NMIBC. Participants will be evaluated for safety and response to AU-011 up to 12 months from initiation of treatment.
  Interventions: Combination Product: AU-011 in Combination with Medical Laser Administration
- Focal injection of AU-011 and laser application with option for TURBT (4e) (Experimental): Participants with intermediate-risk NMIBC will receive multiple treatment cycles of focal AU-011 (400 µg per lesion) followed by laser activation, with the option for TURBT. Participants will be evaluated for safety and response to AU-011 for up to 12 months from initiation of treatment. Enrollment will occur in parallel with Cohort 4g, with randomized (1:1) assignment.
  Interventions: Combination Product: AU-011 in Combination with Medical Laser Administration
- Focal injection of AU-011 and laser application with mandatory TURBT (4f) (Experimental): Participants with high-risk NMIBC will receive multiple treatment cycles of focal AU-011 (400 µg per lesion) followed by laser activation prior to mandatory TURBT. Participants will be evaluated for safety and response to AU-011 for up to 12 months from initiation of treatment.
  Interventions: Combination Product: AU-011 in Combination with Medical Laser Administration
- Focal injection of AU-011 and laser application with optional TURBT (4g) (Experimental): Participants with intermediate-risk NMIBC will receive multiple treatment cycles of focal AU-011 (400 µg per lesion) followed by laser activation with the option of TURBT. Participants will be evaluated for safety and response to AU-011 for up to 12 months from initiation of treatment. Enrollment will occur in parallel with Cohort 4e, with randomized (1:1) assignment.
  Interventions: Combination Product: AU-011 in Combination with Medical Laser Administration
- Focal injection of AU-011 and laser application with option for TURBT (4h) (Experimental): Participants with intermediate-risk NMIBC will receive multiple treatment cycles of focal AU-011 (800 ug per lesion) with laser treatment and option for TURBT. Participants will be evaluated for safety and response to AU-011 up to 12 months from initiation of treatment. This arm is optional and will be run at the discretion of the sponsor.
  Interventions: Combination Product: AU-011 in Combination with Medical Laser Administration
- Focal injection of AU-011 and laser application with mandatory TURBT (4i) (Experimental): Participants with high-risk NMIBC will receive multiple treatment cycles of focal AU-011 (800 µg per lesion) before mandatory TURBT. Participants will be evaluated for safety and response to AU-011 up to 12 months from initiation of treatment. This arm is optional and will be run at the discretion of the sponsor.
  Interventions: Combination Product: AU-011 in Combination with Medical Laser Administration

INTERVENTIONS:
Drug: AU-011 — Administration of AU-011 intratumorally and intramurally
  Arms: Focal injections of AU-011 prior to TURBT (1b)
Combination Product: AU-011 in Combination with Medical Laser Adminstration — AU-011 Intratumorally and Intramurally
  Arms: Focal injections of AU-011 with laser application before TURBT (4a)
Combination Product: AU-011 in Combination with Medical Laser Administration — AU-011 Intratumorally
  Arms: Focal injection of AU-011 and laser application with mandatory TURBT (4f); Focal injection of AU-011 and laser application with mandatory TURBT (4i); Focal injection of AU-011 and laser application with option for TURBT (4d); Focal injection of AU-011 and laser application with option for TURBT (4e); Focal injection of AU-011 and laser application with option for TURBT (4h); Focal injection of AU-011 and laser application with optional TURBT (4g); Focal injection of AU-011 with laser application before TURBT (4b); Focal injection of AU-011 with laser application before TURBT (4c)

SUMMARY:
The main objectives of this study are to determine the feasibility and safety of Belzupacap Sarotalocan (AU-011, bel-sar) treatment of bladder cancer utilizing focal injections with or without laser application.

DETAILED DESCRIPTION:
Aura is enrolling participants with urothelial carcinoma to evaluate the safety, technical feasibility, and preliminary efficacy of bel-sar. The goal is to achieve the trial objectives with minimal disruption to the standard of care (SoC) of the treating Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the following histopathologic requirements for urothelial carcinoma:

   * For Cohorts 1b, 4a-c:

   histopathological diagnosis of NMIBC (any grade) is required. For participants with first diagnosis of NMIBC, confirmation of urothelial carcinoma by recent biopsy (≤6 months of Screening Visit) is required. Participants with recurrent NMIBC must have a current lesion that clinically appears to be NMIBC with histopathologic confirmation based on TURBT or biopsy within the last 24 months).

   For Cohorts 4d, 4e, 4g and 4h, a diagnosis of LG IR NMIBC (according to

   AUA risk classification guidelines) is required, specifically:
   * Multifocal LG Ta; OR
   * Solitary LG Ta >3 cm; OR
   * Low-grade Ta with prior recurrence(s) within 1 year.

   For Cohorts 4f and 4i, a diagnosis of HR NMIBC (according to AUA risk classification guidelines) is required, specifically:
   * Ta HG papillary disease with or without CIS; OR
   * T1 papillary disease with or without CIS
   * Participants may be BCG-naïve or may have received prior treatment with BCG for HR or IR NMIBC (BCG-exposed, BCG-failed, BCG-intolerant)
   * BCG-refractory participants are excluded. BCG-refractory is defined by the following:

     * Persistent HG disease at 6 months following adequate BCG (defined as ≥5/6 induction instillations and ≥2 additional doses, either from re-induction or maintenance), OR
     * HG T1 disease at first evaluation (3 months) after BCG, OR
     * Persistent CIS that remains despite a second BCG course, OR
     * Disease progression in stage or grade during BCG therapy, including maintenance
2. Have no evidence of current or prior metastatic urothelial carcinoma
3. Adequate bone marrow, renal, and hepatic function

Exclusion Criteria:

1. Any additional malignancy that requires active treatment, unless deemed appropriate after discussion by the Investigator with the trial's Medical Monitor.
2. Used an investigational drug or medical device within 30 days or 5 half-lives (whichever is longer) of Visit 1 or be concurrently enrolled in another investigational trial.
3. Active bacterial, fungal, or viral infections - all prior infections must have resolved following optimal therapy and subject must be off all systemic anti-infective agents.
4. Active autoimmune disease, chronic inflammatory condition, or other conditions (like solid organ transplant or bone marrow allograft) requiring concurrent use of any systemic immunosuppressants or steroids.
5. Chronic active hepatitis B or C and HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Safety of AU-011: Incidences of SAEs and DLTs | up to 12 months
  Incidence and severity of treatment-related adverse events [time frame 12 months], serious adverse events [time frame 12 months], and incidence of dose-limiting toxicities [time frame 14 days]

SECONDARY OUTCOMES:
Complete response (CR) rate | at the 3-month time point and at TURBT
  for all cohorts
Duration of response (DoR) | 12 months
  In participants who achieve CR
Durable CR rate | 6-, 9-, and 12-month follow-up
  Proportion of participants maintaining a CR after achieving a CR
Recurrence-free survival (RFS) | 12 mos
  Participants in neoadjuvant cohorts

CONTACTS AND LOCATIONS:
Locations (17):
- United States (11):
  - Arkansas Urology, Little Rock, Arkansas
  - Tower Urology, Los Angeles, California
  - Saint John's Cancer Institute, Santa Monica, California
  - Montefiore Medical Center, The Bronx, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas San Antonio, San Antonio, Texas
  - Urology San Antonio/USA Clinical Trials, San Antonio, Texas
  - The Urology Place, San Antonio, Texas
- Australia (6):
  - Westmead Private Hospital, Westmead, New South Wales
  - Austin Health, Heidelberg, Victoria
  - Warringal Private Hospital, Heidelberg, Victoria
  - Penninsula Private Hospital, Langwarrin, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Hollywood Private Hospital, Nedlands, Washington

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR